CLINICAL TRIAL: NCT07366281
Title: Post-operative Use of the New Adhesive After Total Laryngectomy
Brief Title: Post-operative Use of New Adhesive After Total Laryngectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL_Adhesive
Record Dates: First submitted 2025-12-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Laryngectomy
Keywords: Adhesive baseplate; Tracheostoma care; Postoperative stoma management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploratory post-operative use of Comfort Adhesive (Experimental): Participants will start using a newly developed adhesive called Provox Life Comfort Adhesive in the immediate post-operative period following total laryngectomy.
  Interventions: Device: Provox Life Comfort Adhesive

INTERVENTIONS:
Device: Provox Life Comfort Adhesive — The new Provox Life Comfort adhesive is a medical adhesive baseplate designed for tracheostoma care in laryngectomy patients.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, safety, and performance of the new adhesive when used in the immediate post-operative period after total laryngectomy.

The main question it aims to answer is:

- Is the adhesive feasible and safe to use during the early post-operative phase?

This is a single-arm feasibility study with historical controls, so there is no concurrent comparison group. Researchers will compare outcomes to historical data from standard adhesive use to assess improvements in tolerance and skin condition.

Participants will:

* Use the adhesive as part of their standard post-laryngectomy care.
* Complete patient-reported outcome questionnaires (e.g., comfort, skin assessment, satisfaction).
* Allow investigators to record observations in diaries and patient charts.
* Participate in routine clinical assessments during hospitalization and at end of study (approximately 30 days post-surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing total laryngectomy surgery
* 18 years or older

Exclusion Criteria:

* Unable to give informed consent prior to TL surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Able to Use New Adhesive During Postoperative Period | From enrollment to the end of treatment at 30 days.
  Ability to use new adhesive continuously during the postoperative period, without discontinuation due to intolerance or complications related to the adhesive. Assessed through patient diary and investigator review.

SECONDARY OUTCOMES:
Number of Skin Reactions or Pain/Discomfort Assessed by Investigator and Patient | From enrollment to the end of treatment at 30 days.
  Presence of skin reactions under or around the adhesive and pain/discomfort, assessed by investigator and patient. Skin condition evaluated using the Skin Integrity Severity Assessment Scale (0 = Normal, 1 = Mild, 2 = Moderate, 3 = Severe) and investigator assessment of erythema, vesicles, maceration, skin tears, crusting, and edema. Includes reported discomfort (VAS 0-10).
Performance: Adhesive Adhesion Performance: Score on 5-Point Adhesion Rating Scale | From enrollment to the end of treatment at 30 days.
  Ability of adhesive to remain attached during intended wear period, assessed on a 5-point scale of Adhesion Rating Scale, that ranges from "Adhesion of Adhesive is very bad " to "Adhesion of Adhesive is very good".
Device Life Measured as Hours Adhesive Remains in Place | From enrollment to the end of treatment at 30 days.
  Hours adhesive remains in place before replacement.
Performance: Adequacy of Adhesive Fit Around Stoma on a 5-Point Stoma Fit Scale | From enrollment to the end of treatment at 30 days.
  Investigator and patients assessment of adhesive fit around stoma, assessed on a 5-point Stoma Fit scale ranging from "Adhesive does not fit at all" to "Adhesive fits very well".
Performance: Ease of Adhesive Application and Removal on 5-Point Ease Scale | From enrollment to the end of treatment at 30 days.
  Patient and investigator rating/assessment of how easy adhesive is to apply and remove, assessed on a 5-point scale ranging from "Very difficult" to "Very easy".
Performance: Ability to Observe Area Underneath Adhesive | From enrollment to the end of treatment at 30 days.
  Whether skin under adhesive can be inspected without removal.
Number of Participants for Whom Adhesive Was Successfully Applied Directly Over Sutures Without Complications | From enrollment to the end of treatment at 30 days.
  Feasibility of applying adhesive over sutures without complications.
Number of Participants Able to Speak Using the Comfort Adhesive | From enrollment to the end of treatment at 30 days.
  Ability to speak while the Comfort Adhesive is in place will be assessed by both the patient and the investigator using a binary response (Yes/No). A "Yes" response indicates the participant is able to speak with a voice prosthesis while using the Comfort Adhesive. Higher frequency of "Yes" responses reflects a better outcome.
Pulmonary rehabilitation: Average Hours of Heat and Moisture Exchanger Use per 24 Hours | From enrollment to the end of treatment at 30 days.
  Hours of heat and moisture exchanger use per 24 hours.
Pulmonary rehabilitation: Interference With Sputum Clearance While Using Adhesive: Score on 4-Point Mucus Trapping Scale | From enrollment to the end of treatment at 30 days.
  Difficulty with sputum clearance while using the adhesive will be assessed by patient and investigator using a 4-point Mucus Trapping Scale ranging from "Mucus gets often trapped under the adhesive" to "Mucus never gets trapped under the adhesive".
Use of Supplemental Oxygen During Postoperative Period | From enrollment to the end of treatment at 30 days.
  Need for supplemental oxygen will be assessed by investigator confirmation using a categorical response:
  * Yes (used supplemental oxygen throughout)
  * Yes, but weaned (used initially, then discontinued)
  * No (did not use supplemental oxygen)
Patient-Reported Comfort Level: Score on 5-Point Comfort Scale | From enrollment to the end of treatment at 30 days.
  Patient-reported comfort level using adhesive, assessed on a 5-point Comfort Scale ranging from "Very Uncomfortable" to "Very Comfortable."

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No